CLINICAL TRIAL: NCT00578578
Title: Protocol for a Randomized, Placebo-Controlled, Double-Blinded Trial to Study the Effects of Supplementary Omega-3 Fatty Acids on Serum C-Reactive Protein Levels
Brief Title: Trial to Study the Effects of Supplementary Omega-3 on Serum C-Reactive Protein Levels
Acronym: Omega-3
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: CRP is no longer SOC - enrollment halted and will analyze available data.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Deepak Bhatt, MD, Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB# 6970; IRB# 6970
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Coronary Artery Disease; Inflammatory Response; Atherosclerosis
Keywords: Omega3 fatty acids; hsCRP; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active Arm:
  1000 mg Lemon flavored Capsules. Three capsules every morning.
  Interventions: Dietary Supplement: eicosapentaenoic acid (EPA),
- 2 (Placebo Comparator): Placebo Arm:
  Cornstarch Capsules provided by Clinical Encapsulation services. Three capsules every morning.
  Interventions: Dietary Supplement: eicosapentaenoic acid (EPA),

INTERVENTIONS:
Dietary Supplement: eicosapentaenoic acid (EPA), — three capsules daily (1350 mg daily) of EPA for 8 weeks or three capsules daily placebo for 8 weeks
  Other Names: Omega 3

SUMMARY:
To study the anti-inflammatory effects of marine omega-3 fatty acids, also known as n-3 polyunsaturated fatty acids (PUFA), we propose a randomized, double-blinded, prospective, single-center trial to examine the effect of supplementary n-3 PUFA on serum high sensitivity (hs) CRP levels.

Inclusion Criteria Age > 18 hs CRP >3mg/L and <10 mg/L

Exclusion Criteria

Active infection Systemic Inflammatory Disease Autoimmune disorders Systemic Lupus Erythematosus (SLE) Rheumatoid Arthritis (RA) Systemic Sclerosis (Scleroderma) Sjögren's Syndrome Behçet's Syndrome

The Vasculitis Syndromes Including:

Wegener's granulomatosis Temporal arteritis (Giant cell arteritis) Takayasu's arteritis Henoch-Schönlein purpura Predominantly cutaneous vasculitis (hypersensitivity vasculitis) Sarcoidosis Amyloidosis Currently on warfarin Cr > 2.0 Fish Allergy Pregnancy or unwillingness to use some form of birth control in women of child-bearing age during the 8 weeks.

We will enroll 200 pts. at Willoughby Hills Family Health Center over a 2 month period 100 pts. will receive OMEGA-3, 100 pts. will receive placebo Drug is to be taken over 8 weeks Pt. will return to Willoughby Hills in 8 weeks for a follow-up hsCRP. A brief questionnaire will be completed by the nurse/pt, including vital signs at baseline and follow-up .

Primary Outcome:

hsCRP levels after 8 weeks of treatment with PUFA

DETAILED DESCRIPTION:
All patients will be given an 8 week supply of placebo or study drug. The exact composition of both the active drug and placebo is detailed below. The physician and the patient will both be blinded. Patients will be instructed to take three capsules daily in the morning. Each capsule of the drug contains 450 mg of eicosapentaenoic acid (EPA), the active component. Thus, three capsules daily will result in 1350 mg daily of EPA. They will be asked to return to the clinic after 8 weeks of therapy for a follow-up hsCRP.

Patients:

Healthy patients seen in a primary care setting at the Department of Internal Medicine at the Cleveland Clinic Health System Willoughby satellite.

Drug:

Active Arm:

1000 mg Lemon flavored Capsules. Three capsules every morning.

Fill

45% Eicosapentaenoic Acid 10% Docosahexaenoic Acid 10% Combined total of Docopentaneoic Acid and Alfa-Linoleic Acid Natural Lemon Oil Rosemary Liquid Extract D-alpha Tocopherol Vitamin E (67.1% W/W) (1000IU/G) Antioxidants, proprietary mix

Shell

Gelatin Glycerol Purified Water Lemon Oil

Placebo Arm:

Cornstarch Capsules provided by Clinical Encapsulation services. Three capsules every morning.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* hs CRP >3mg/L and <10 mg/L

Exclusion Criteria:

* Active infection
* Systemic Inflammatory Disease
* Currently on warfarin
* Cr > 2.0
* Fish Allergy
* Pregnancy or unwillingness to use some form of birth control

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
hsCRP levels after 8 weeks of treatment with PUFA | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Bhatt, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Willoughby Hills Family Health Center, Willoughby Hills, Ohio, United States